CLINICAL TRIAL: NCT00728416
Title: Placebo-Controlled Study of Mometasone Furoate Nasal Spray (MFNS) 200 mcg QD in the Relief of Nasal Congestion Associated With Seasonal Allergic Rhinitis (SAR)
Brief Title: Study of Nasonex in the Relief of Nasal Congestion in Patients With Seasonal Allergic Rhinitis (Study P05583)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05583; MK-0887-160 (Other: Merck)
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Mometasone furoate nasal spray 200 mcg QD (once per day)
  Interventions: Drug: Mometasone furoate nasal spray (MFNS)
- Arm 2 (Placebo Comparator): Matching placebo nasal spray
  Interventions: Drug: Matching placebo nasal spray

INTERVENTIONS:
Drug: Mometasone furoate nasal spray (MFNS) — MFNS 50 mcg/spray: two sprays in each nostril once daily (ie, 200 mcg QD) for 15 days
  Other Names: MK-0887, Nasonex Nasal Spray
  Arms: Arm 1
Drug: Matching placebo nasal spray — Matching placebo nasal spray: 2 sprays in each nostril once daily for 15 days
  Other Names: Placebo
  Arms: Arm 2

SUMMARY:
This study seeks to prospectively demonstrate that Nasonex is better than placebo in relieving nasal congestion in patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be 12 years of age or older, of either sex, and of any race.
* A subject must have at least a 2-year history of SAR which exacerbates during the study season.
* A subject must have a positive skin prick test response to an appropriate seasonal allergen at Visit 1.
* A subject must be clinically symptomatic at the Screening and Baseline Visits.

Exclusion Criteria:

* A subject with a history of severe local reaction(s) or anaphylaxis to skin testing.
* A subject who has had an upper respiratory tract or sinus infection that required antibiotic therapy without at least a 14-day washout prior to the Screening Visit, or who has had a viral upper respiratory infection within 7 days prior to the Screening Visit.
* A subject who has used any drug in an investigational protocol in the 30 days prior to the Screening Visit.
* A subject who is participating in any other clinical study.
* A subject who is part of the staff personnel directly involved with this study.
* A subject who is a family member (parent, spouse, or sibling) of the investigational study staff.
* A female subject who is breast-feeding, pregnant, or intends to become pregnant.
* A subject previously randomized into this study.
* A subject who has a family member (parent, spouse, or sibling) currently enrolled in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Meltzer EO, Shekar T, Teper AA. Mometasone furoate nasal spray for moderate-to-severe nasal congestion in subjects with seasonal allergic rhinitis. Allergy Asthma Proc. 2011 Mar-Apr;32(2):159-67. doi: 10.2500/aap.2011.32.3424. PMID 21439168

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray: Mometasone furoate nasal spray 200 mcg QD (once per day)
- Placebo Nasal Spray: Matching placebo nasal spray
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 168 | 165
Completed | 166 | 163
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Treatment Failure | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 168 | 165 | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 148 | 146 | 294
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 103 | 212
  Male | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM/PM PRIOR Nasal Congestion Score Over 15 Days
Description: Nasal congestion was scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. PRIOR (the subject's status over the previous 12 hours [reflective]). Baseline is the average score from the 3 days prior to the first dose of study drug.
Time Frame: 15 days of treatment
Population: 1 participant without baseline value excluded from the Placebo Nasal Spray population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 168 | 164
Units on a scale | -0.71 (0.55) [-0.81 to -0.61] | -0.40 (0.55) [-0.50 to -0.30]
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; The change from Baseline in average AM/PM PRIOR nasal congestion score over 15 days: MFNS 200 mcg daily vs placebo. The difference in LS means (MFNS - Placebo) was calculated from an ANCOVA model with treatment, site and baseline AM/PM PRIOR Nasal Congestion Score as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LS Means = -0.31, 95% CI 2-sided [-0.43 to -0.19]

2. Secondary Outcome: Change From Baseline in Average AM/PM PRIOR Total Nasal Symptom Score Over 15 Days
Description: Total nasal symptom score (TNSS) is a composite of 4 symptoms, each is scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total can range from 0 to 12. PRIOR (the subject's status over the previous 12 hours [reflective]). Baseline is the average score from the 3 days prior to the first dose of study drug.
Time Frame: 15 days of treatment
Population: 1 participant without baseline value excluded from the Placebo Nasal Spray population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 168 | 164
Units on a scale | -3.00 (2.03) [-3.38 to -2.62] | -1.73 (2.03) [-2.11 to -1.34]
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; The change from Baseline in average AM/PM PRIOR TNSS over 15 days: MFNS 200 mcg daily vs placebo. The difference in LS means (MFNS - Placebo) was calculated from an ANCOVA model with treatment, site and baseline AM/PM TNSS as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LS Means = -1.27, 95% CI 2-sided [-1.72 to -0.83]

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after study completion/discontinuation (up to 45 days)
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/165
Other Adverse Events (participants affected / at risk) | 0/168 | 0/165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days